CLINICAL TRIAL: NCT04636424
Title: Weight Distribution Asymmetry in Relation to Speed During Gait in Children With Spastic Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ibrahim, Doctoral degree (lecturer), Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: correlation study
Record Dates: First submitted 2020-11-08; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gait, Spastic
Keywords: assymetry-gait-speed-cerebral palsy
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spastic diplegic group (Experimental): assessment of the speed and weight distribution during gait
  Interventions: Other: assesment of gait
- hemiplegic group (Experimental): assessment of the speed and weight distribution during gait
  Interventions: Other: assesment of gait

INTERVENTIONS:
Other: assesment of gait — speed and weight distribution during gait

SUMMARY:
Background: Improving walking ability is one of the major concerns in therapeutic interventions for children with cerebral palsy.

Aim: determine the relation between the weight distributed on both lower limb and speed during walking.

DETAILED DESCRIPTION:
sixty children with spastic diplegia (group A) and forty-five with hemiparesis ( group B) with age ranged from ten to twelve, they had spasticity grade 1 and 1+ according to modified ashworth scale and they were able to walk with assistance (level II on Gross Motor Classification System).Evaluation was held by the Biodex gait trainer for measuring weight distribution on both lower limbs and speed during gait to determine if there was a relation between weight distribution asymmetry and the speed of gait of those children

ELIGIBILITY:
Inclusion Criteria:

The selection criteria to the diplegic group were as follows:

1. children diagnosed as spastic diplegia or hemiplegia;
2. the ability to stand independently without support for not less than 30 seconds;
3. the ability to walk independently; a classification of level II in the Gross Motor Function Classification System (GMFCS);
4. and capability to understand simple verbal commands.

Exclusion criteria:

1. Participants were excluded if they were treated for lower limbs orthopedic surgical or with botulinum toxin injection within the last 6 months
2. or if they had fixed lower limb deformity.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
speed of gait | 12 weaks
  the velocity of walking

SECONDARY OUTCOMES:
foot to foot distribution | 12 weaks
  weight loaded on each lower limb during gait assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Mohamed, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy,Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the results will be shared with other researchers as the paper published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication of the paper
Access Criteria: through the journal of the published paper

REFERENCES:
- [Background] Nahla M. Ibrahim, Mai Elsayed Abbass. EFFECT OF PEDAL TRAINING ON GAIT SPEED IN CHILDREN WITH HEMIPARETIC CEREBRAL PALSY.Int J Physiother Res 2017;5(6):2560-65. ISSN 2321-1822